CLINICAL TRIAL: NCT04607551
Title: PRONing to Facilitate Weaning From ECMO in Patients With Refractory Acute Respiratory Distress Syndrome
Acronym: PRONECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP180607; 2019-A02669-48 (Other: IDRCB)
Record Dates: First submitted 2020-09-28; First posted 2020-10-29 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-06

CONDITIONS: ARDS
Keywords: ECMO Weaning; PRONING
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone positionning (Experimental)
  Interventions: Procedure: Prone positionning
- Supine position (Active Comparator)
  Interventions: Procedure: Supine position

INTERVENTIONS:
Procedure: Prone positionning — 4 to 5 persons required for the procedure, one of them being dedicated to the management of the head of the patient, the endotracheal tube, the jugular ECMO cannula and the ventilator lines and another dedicated to the femoral ECMO cannula. The person at the head of the bed will coordinate the steps. The other persons will stand at each side of the bed. The direction of the rotation will be decided giving priority to the side of the central venous lines. The length of vascular and ventilator lines will be checked for appropriateness, the endotracheal tube and gastric tube will be secured, and the patient's knees, forehead, chest, and iliac crests will be protected using adhesive pads. The patient will be then moved along the horizontal plane to the opposite side of the bed selected for the direction of rotation. Patients will be proned at least four times during the first days on ECMO. Each prone session will stand for at least 16 hours
  Arms: Prone positionning
Procedure: Supine position — Patients assigned to supine will remain in a semi-recumbent position.
  Arms: Supine position

SUMMARY:
ECMO has emerged as a promising intervention that may provide more efficacious supportive care to patients with refractory severe acute respiratory distress syndrome (ARDS). The largest randomized trial of ECMO for severe forms of ARDS was recently published and demonstrated no significant benefit from early initiation of ECMO with respect to 60-day mortality, when compared with a strategy of conventional mechanical ventilation (MV) (ref EOLIA). However, a rescue ECMO option was used by 28% of the controls, which is likely to have diluted the potential positive effect of ECMO. One may argue that a less restrictive primary endpoint, such as death or rescue ECMO, would have yielded positive findings.

Meanwhile, improvements in technology have made ECMO safer and easier to use, allowing for the potential of more widespread application in patients with ARDS. VV-ECMO can be used as a life-saving rescue therapy in patients with ARDS when MV cannot maintain adequate oxygenation or CO2 elimination. Alternatively, VV-ECMO may be used in patients who remain hypoxemic during MV (i.e., PaO2/FiO2<80 mmHg) despite optimization of MV (including the application of high levels of positive end-expiratory pressure (PEEP), neuromuscular blockers, and prone positioning) and allow "lung rest" by lowering airway pressures and tidal volume to ameliorate ventilator-induced lung injury (VILI).

Prone positioning (PP) has been used for more than 30 years in patients with acute hypoxemic respiratory failure and in particular with ARDS. Initially, PP in ARDS patients was proposed as an efficient mean to improve oxygenation, sometimes dramatically, in a large number of patients. In addition, it is now clear, and data are still accumulating, that PP is also able to prevent VILI which is as important as maintaining safe gas exchange in mechanical ventilation. Therefore, PP is a strategy that covers the two major goals of ventilator support in ARDS patients, maintaining safe oxygenation and preventing VILI and reducing mortality at the end. This latter objective makes sense on ECMO as one of the main objective of this device is to markedly reduce VILI by resting the lung.

Considering that PP is a valuable and safe therapy to reduce VILI, its combination with ECMO could enhance VILI prevention. In recent preliminary studies, it was reported that the combination of VV-ECMO and PP was associated with a dramatic improvement in oxygenation, in pulmonary and thoracic compliance and in chest X-ray findings. It may thus facilitate the weaning of ECMO and can be performed without compromising the safety of the patients. Lung recruitment and improvement in ventilation/perfusion mismatch on prone position may both contribute to improve oxygenation. PP may therefore be efficient to hasten the weaning of VV-ECMO when atelectasis and ventilation/perfusion mismatch occur under ultra-protective ventilation even in patients in whom pre-ECMO PP failed. In addition, it could also enhance ventilator induced lung injury prevention on ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. Severe ARDS refractory to conventional therapy placed on VV-ECMO support in the preceding 48h.
2. Obtain informed consent from a close relative or surrogate. According to the specifications of emergency consent, randomization without the close relative or surrogate consent could be performed.

   Close relative/surrogate/family consent will be asked as soon as possible. The patient will be asked to give his/her consent for the continuation of the trial when his/her condition will allow.
3. Social security registration

Exclusion Criteria:

1. Age <18 and >75
2. Pregnancy and breastfeeding woman
3. Initiation of VV-ECMO >48 h
4. Resuscitation >10 minutes before ECMO
5. Irreversible neurological pathology
6. End-stage chronic lung disease
7. ARDS secondary to an abdominal surgery
8. Contraindications for PP
9. Irreversible ARDS with no hope for lung function recovery
10. Patient moribund on the day of randomization, SAPS II >90
11. Liver cirrhosis (Child B or C)
12. Chronic renal failure requiring hemodialysis
13. Lung transplantation
14. Burns on more than 20 % of the body surface

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Time to successful ECMO weaning within the 60 days following randomization | Day 60
  ECMO weaning will be considered successful only if the patient survives without ECMO, or lung transplantation 30 days after ECMO removal. Thus all ECMO weaning from randomization to 60 days after randomization will be considered, and the qualification for successful ECMO weaning will need 30 days of follow-up after ECMO removal (thus until day 90 after randomization for an ECMO weaning performed on day 60 after randomization).
  Patients still under ECMO 60 days after randomization will be censored.
  A protocolized management regarding weaning of VV-ECMO will be applied to both groups
  The planned analysis will model the risk of successful ECMO ablation in the presence of competing risk (death and weaning failure).

SECONDARY OUTCOMES:
Mortality | Day 7, Day 14, Day 30, Day 60, Day 90
Total duration of ECMO support | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90,
Number of ECMO-free days | Between day 1 and Day 60/Day 90
Duration of ICU stay | Between day 1 and Day 60/Day 90
Duration of hospitalization | Between day 1 and Day 60/Day 90
Time to improvement in respiratory respiratory system compliance | Through study completion
Time to get a respiratory system compliance > 30 mL/cmH2O | Between day 1 and Day 60/Day 90
Number of days with organ failure | Between day 1 and Day 60
  defined by SOFA score
Number of days alive without organ failure | Between day 1 and Day 60
  defined by SOFA score
Number of ventilator assist pneumonia, bacteriemia, and cannula infection episodes | Through study completion
Number of days with hemodynamic support with catecholamines | Between day 1 and Day 60
Number of days alive without hemodynamic support with catecholamines | Between day 1 and Day 60
Number of days with mechanical ventilation | Between day 1 and Day 60
Number of days alive without mechanical ventilation | Between day 1 and Day 60
Acute core pulmonale diagnosis | Between day 1 and D60
  by echocardiography
Need for VA ECMO | Between day 1 and Day 60/Day 90
Incidence of intervention side effects | Between day 1 and Day 60
  (accidental decannulation, non-scheduled extubation during the procedure, hemoptysis, endotracheal tube obstruction, cardiac arrest, pressure sore, and death
Occurrence of refractory hypoxemia on ECMO | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Schmidt M, Hajage D, Lebreton G, Dres M, Guervilly C, Richard JC, Sonneville R, Winiszewski H, Muller G, Beduneau G, Mercier E, Roze H, Lesouhaitier M, Terzi N, Thille AW, Laurent I, Kimmoun A, Combes A; PRONECMO Investigators, the REVA Network, and the International ECMO Network (ECMONet). Prone Positioning During Extracorporeal Membrane Oxygenation in Patients With Severe ARDS: The PRONECMO Randomized Clinical Trial. JAMA. 2023 Dec 26;330(24):2343-2353. doi: 10.1001/jama.2023.24491. PMID 38038395